CLINICAL TRIAL: NCT02270671
Title: Attention Bias Modification Training for Socially Anxious Adolescents: A Randomized Control Trial
Brief Title: Attention Bias Modification Training for Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Amanda Fitzgerald, Lecturer, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-14-49-Fitzgerald
Record Dates: First submitted 2014-10-09; First posted 2014-10-21 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Anxiety; Depression
Keywords: Social Anxiety; Social Phobia; Depression; Attention Bias Modification Training
MeSH Terms: conditions — Anxiety Disorders; Depression; Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo protocol consists of 160 trials (120 angry-neutral face pair and 40 neutral-neutral face pair presentations). In this condition, angry-face location, probe location and actor are fully counterbalanced in presentation. A short break is delivered every 40 trials (1 block). An accuracy of 70% or above for each block is necessary to continue training. The task takes 7 minutes.
  Interventions: Other: Placebo
- Intervention (Experimental): The attention bias modification training (ABMT) protocol consists of 160 trials (120 angry-neutral face pair presentations and 40 neutral-neutral face pair presentations). In the ABM condition, the target-probe appears at the neutral-face locations in all angry-neutral trials. A short break is delivered every 40 trials (1 block). An accuracy of 70% or above for each block is necessary to continue training. The task takes 7 minutes.
  Interventions: Behavioral: ABMT

INTERVENTIONS:
Behavioral: ABMT — Attention Bias Modification Training
  Arms: Intervention
Other: Placebo — Placebo Training
  Arms: Placebo

SUMMARY:
Attention bias modification training (ABMT) is a computer-based attention training programme designed to modify the way a person's attention is directed to mild threats in the environment. What a person focuses their attention on plays an important role in how safe or unsafe they feel in certain situations. Much research has shown that people with high levels of anxiety tend to focus their attention on negative information in their surroundings. The purpose of ABMT is to set in place attention patterns that do not lead to excessive anxiety. The present study will test whether this treatment is effective in reducing social anxiety in 15-18 year olds in school settings.

The study design consists of two phases. During Phase 1 participants will complete a screening questionnaire in relation to their wellbeing and emotions. This questionnaire will include a measure of the affective, cognitive, and behavioural components of social anxiety in adolescence. Depending on their suitability (i.e. scoring above a cut-off on a standardised measure of social anxiety in Phase 1 of the study), participants may then be invited to take part in a 4-week computer-based attention training programme. The purpose of this phase is to see if ABMT will help young people feel less worried or nervous in social situations by teaching them to focus on their environment differently.

Previous research containing attention training tasks similar to this training programme suggests that attention training can reduce symptoms of social anxiety in adolescents. Individuals who are invited to take part in the training session will be randomly assigned to either the intervention (ABMT) or placebo (inactive) group. Both groups will be asked to complete a 4-week programme involving one computer training session per week (each session takes approximately 15-20 minutes).

Questionnaires will also be given to participants to complete before and after the intervention, along with a 12-week follow up assessment. These will include questionnaires to measure social anxiety, depressive symptoms, and fears in relation to negative evaluation. Each questionnaire will take approximately 40 minutes to complete. Participants will not know whether they have received the intervention or placebo training until after the intervention.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is among the most prevalent mental disorders in adolescence (Merikangas et al., 2010), 10% of females and 5% of males are diagnosed with SAD in adolescence (Wittchen & Fehm, 2003). SAD is characterised by marked fear or anxiety about social situations in which the individual is exposed to possible scrutiny by others (APA, 2013). SAD is associated with social isolation, poor social skills, low self-esteem, and future comorbid mental disorders (Wittchen et al., 2000). Social anxiety typically develops during adolescence, thus there is a need to detect and treat it early prior to the development of a clinically-diagnosed SAD. Most early interventions for social anxiety have used Cognitive Behavioural Therapy (CBT), which focuses on modifying explicit verbal cognitions (Neil & Christensen, 2009). However, many adolescents do not have access to CBT and many finding it demanding (Otto et al., 2004).

Recently, researchers have developed a novel treatment, Attention Bias Modification (ABM), which aims to modify implicit cognitive biases (MacLeod, 2012). ABM is based on cognitive theories, which propose that individuals with anxiety automatically attend to threat-related information in their environment, and have a bias towards negative information. In support of these theories, research demonstrates a relationship between attention and anxiety (Mathews & MacLeod, 2002), and this relationship appears to be causal (Mogg & Bradley, 1998). Evidence indicates that social anxiety can be reduced through ABM procedures in clinical (Amir et al., 2008) and non-clinical populations (Klump & Amir, 2009). However, little ABM research has been conducted with adolescents (Sportel et al., 2013). Beard et al. (2011) noted that few ABM studies followed the Consolidated Standards of Reporting Trials guidelines, and few have registered as clinical trials (Emmelkamp, 2012).

The Present Study:

This research tests the efficacy of ABM training in reducing social anxiety in adolescents. Given that the age of onset of social anxiety is adolescence, peaking in late teens (Merikangas et al., 2010), this research focuses on 15-18 year olds. Given that no published study has specifically considered the role of gender and its impact on ABM training, this research builds gender into the design, thus the research is in line with best practice (EU Commission, 2011).

Aims & Objectives:

1. To test the efficacy of ABM training in reducing social anxiety in adolescents
2. To examine the impact of gender on the efficacy of ABM training in reducing social anxiety

Central Research Questions:

1. Is ABM training associated with:

   I. A decrease in threat-related attentional biases? II. A decrease in negative evaluations? III. A decrease in social anxiety? IV. A decrease in test anxiety?
2. Does gender have an impact on the efficacy of ABM in reducing social anxiety?

PHASE 1: PRE-SCREEN FOR SOCIAL ANXIETY IN ADOLESCENTS Objective: To screen for sub-clinical levels of social anxiety in adolescents.

School Sampling: 4-8 large second-level schools in Dublin will be randomly selected from the Department of Education and Skills 2012 published list of schools. Schools will be gender-mixed and matched for school size, disadvantaged/non-disadvantaged status, and geographical location.

Power Analysis: Using G*Power 3.1, the sample size was determined as 80 based on the following parameters: a medium effect size of 0.3, alpha of 0.05, power of 0.8, a repeated measures within-between interaction: 2 (Group: ABM, Placebo) X 2 (Gender: Female, Male) X 3 (Time: Pre, Post, Follow-up). To account for attrition rates, a sample of 100 participants will be recruited.

Participants: Adolescents aged 15-18 years in Senior Cycle will be invited for the initial screening.

Procedure: Adolescents must return parental and informed consent forms. Participants will be screened using the Social Phobia and Anxiety Inventory for Children (SPAI-C, Beidel et al., 1998). Participants scoring above the cut-off for social anxiety on the SPAI-C will be invited to participate in the intervention (Phase 2).

Approximately, 1500 Senior Cycle students across 8 schools will be invited to complete the pre-screen in Phase 1. With an approximate response rate of 50% (N=500), and using the 25% top centile a sample of 125 will be identified. Because of anticipated drop-out, the investigators will randomly select 100 adolescents for the intervention (50 per condition).

PHASE 2: RANDOMIZED CONTROL TRIAL Objective: To compare the efficacy of ABM to placebo training in reducing social anxiety.

Participants: Adolescents from Phase 1 screening above cut-off will be invited to participate in the intervention and randomly assigned to the ABM/placebo training. On the basis of pre-screening from Phase 1, the PI will ensure group equivalence across ABM versus placebo group in key variables (e.g., age, gender, social anxiety) in advance of randomization. Post randomization, independent variables will be checked to ensure they are balanced across groups so as not to contaminate outcomes of the study.

Procedure:

ABM and Placebo Protocols Participants in both ABM and placebo training groups will receive 4 training sessions over a 4-week period. The intervention will be performed on a laptop during school and delivered in a quiet room with the researcher present. Pre-test will occur prior to the intervention, post-test will be after 4 weeks, followed by follow-up assessment at 12 weeks.

The Dot-Probe Attention Task The dot-probe task forms the basis for both threat bias assessment and attention bias modification. In the dot-probe task, pairs of faces (stimuli), one threat-related (angry face) and one neutral (neutral face) are presented at different locations on a computer screen at the same time on each trial. Each trial begins with the presentation of a fixation display (500ms; white cross at the centre of the screen), on which the participant is requested to focus their gaze. The fixation display is followed by a face pair display (500ms). Immediately following the face pair display, a target-probe appears. The target-probe consists of an arrowhead pointing either left or right ("<" or ">"), and appears at the location previously occupied by one of the faces. Participants are required to determine which symbol appeared by pressing one of two pre-specified buttons on a mouse. Participants are required to respond as quickly as possible to the target-probe without compromising accuracy. Response latencies on this task provide a 'snap-shot' of the distribution of the participant's attention, with faster responses to target-probes presented in the attended location relative to the unattended location. Attention bias to threat is evident when participants are faster to respond to target-probes that replace threat-related stimuli rather than neutral stimuli. A new trial begins following an inter-trial interval (500ms). The computer training requires E-Prime 2 software (PST, Pittsburgh, PA).

Cue stimuli are face photographs of 20 different individuals (10 male, 10 female) from the NimStim stimulus set (Tottenham, et al., 2009). Two different pictures of each individual are selected, depicting angry and neutral expressions. Participants are presented with pairs of faces of the same actor (neutral face-angry face or neutral face-neutral face) on screen for each trial.

ABM (Intervention) Training The ABM protocol consists of 160 trials (120 angry-neutral face pair presentations and 40 neutral-neutral face pair presentations). In the ABM condition, the target-probe appears at the neutral-face locations in all angry-neutral trials. A short break is delivered every 40 trials (1 block). An accuracy of 70% or above for each block is necessary to continue training. The task takes 7 minutes.

Placebo Training The placebo protocol consists of 160 trials (120 angry-neutral face pair and 40 neutral-neutral face pair presentations). In this condition, angry-face location, probe location and actor are fully counterbalanced in presentation. A short break is delivered every 40 trials (1 block). An accuracy of 70% or above for each block is necessary to continue training. The task takes 7 minutes.

Outcome Measures:

Outcome measure will be administered to all participants in the randomized controlled trial pre-intervention (baseline), post-intervention (week 4), and at 12-week follow-up, including:

Threat Bias Measurement The threat bias measurement protocol consists of 120 trials (80 angry-neutral and 40 neutral-neutral presentations). Angry-face location, probe location, probe type, and actor are fully counterbalanced in presentation. The participant must perform with more than 70% accuracy on the first 10 trials. The task takes 5 minutes.

Social Phobia and Anxiety Inventory for Children (SPAI-C) The SPAI-C (Beidel et al., 1998) is a 26-item self-report instrument and has good psychometric properties with adolescent samples (Inderbitzen-Nolan et al., 2004). The SPAI-C measures the somatic, cognitive and behavioural aspects of social phobia in children and adolescents. Questions relate to how nervous the respondent feels when carrying out certain tasks and response are rated on a 3-point scale from never, or hardly ever to most of the time, or always with higher scores indicating greater levels of social anxiety. In the present study, those participants scoring above the cut-off on the SPAI-C in Phase 1 of the study will be invited to take part in Phase 2 of the study.

Brief Fear of Negative Evaluations Scale - Revised (BFNE-R) Negative evaluations are an important aspect of social anxiety. The BFNE (Carleton et al., 2006) is a 12-item measure which assesses fear of negative evaluation. Items are responded to on a 5-point Likert scale from 0 to 4. The BFNE-R has shown high internal consistency and correlates well with the original BFNE (Carleton et al., 2006).

Screen for Child Anxiety Related Disorders (SCARED) Child Version The SCARED developed by Birmaher et al. (1999) is used to screen for signs of anxiety disorders. The 41-item measure is used to measure anxiety, including panic, separation anxiety, generalised anxiety, social avoidance and school phobia. It has shown high reliability with adolescents (Birmaher et al., 1999). Items are rated on a 3-point Likert scale. Internal consistencies have been shown to be high with adolescent samples (Crocetti et al., 2009).

Depression Subscale of the Revised Child Anxiety and Depression Scale (RCADS) The RCADS (Chorpita et al., 2000) is a 47-item self-report measure and has good psychometric properties with adolescent samples (Mathyssek et al., 2013) The Depression Subscale contains 10 items and will be used in this research. Items relating to the frequency with which depressive symptoms are experienced are rated on a 4-point Likert scale from never to always.

Research Design: A mixed model 2 (Group) x2 (Gender) x3 (Time) complex design combining between subjects and within subjects will be employed. Each participant will be tested at pre-intervention, post-intervention, and follow-up.

Independent Variables:

Group (K=2; ABM/ Placebo) Gender (K=2) Time (K=3; Pre-intervention[baseline], Post-intervention [week 4], and Follow-up)

Analyses:

All analyses on change in social anxiety, anxiety, depression, and fear of negative evaluation will be conducted as intention-to-treat analyses.

1. Descriptive statistics
2. Chi-square analyses and ANOVAs
3. Primary analyses will consist of three-way repeated ANOVAs 2 (Group) x2 (Gender) x3 (Time) to test the variables under study.

ELIGIBILITY:
Inclusion Criteria:

* Those who score above the cut-off on the SPAI-C

Exclusion Criteria:

* Those with a diagnosed mental health disorder
* Those who are currently attending a mental health professional
* Those scoring below the cut-off on the SPAI-C
* Those who decline to participate
* Those whose parents/guardians do not provide written consent

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Fitzgerald, Ph.D., Principal Investigator — University College Dublin; Barbara Dooley, Ph.D., Principal Investigator — University College Dublin; Yair Bar-Haim, Ph.D., Study Chair — Tel Aviv University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wittchen HU, Fehm L. Epidemiology and natural course of social fears and social phobia. Acta Psychiatr Scand Suppl. 2003;(417):4-18. doi: 10.1034/j.1600-0447.108.s417.1.x. PMID 12950432
- [Background] Wittchen HU, Carter RM, Pfister H, Montgomery SA, Kessler RC. Disabilities and quality of life in pure and comorbid generalized anxiety disorder and major depression in a national survey. Int Clin Psychopharmacol. 2000 Nov;15(6):319-28. doi: 10.1097/00004850-200015060-00002. PMID 11110007
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition. Arlington, VA, American Psychiatric Association, 2013.
- [Background] Neil AL, Christensen H. Efficacy and effectiveness of school-based prevention and early intervention programs for anxiety. Clin Psychol Rev. 2009 Apr;29(3):208-15. doi: 10.1016/j.cpr.2009.01.002. Epub 2009 Jan 25. PMID 19232805
- [Background] Otto MW, Smits JA, Reese HE. Cognitive-behavioral therapy for the treatment of anxiety disorders. J Clin Psychiatry. 2004;65 Suppl 5:34-41. PMID 15078117
- [Background] Macleod C. Cognitive bias modification procedures in the management of mental disorders. Curr Opin Psychiatry. 2012 Mar;25(2):114-20. doi: 10.1097/YCO.0b013e32834fda4a. PMID 22227631
- [Background] Mathews A, MacLeod C. Induced processing biases have causal effects on anxiety. Cognition and Emotion 16(3): 331-354, 2002.
- [Background] Mogg K, Bradley BP. A cognitive-motivational analysis of anxiety. Behav Res Ther. 1998 Sep;36(9):809-48. doi: 10.1016/s0005-7967(98)00063-1. PMID 9701859
- [Background] Amir N, Weber G, Beard C, Bomyea J, Taylor CT. The effect of a single-session attention modification program on response to a public-speaking challenge in socially anxious individuals. J Abnorm Psychol. 2008 Nov;117(4):860-868. doi: 10.1037/a0013445. PMID 19025232
- [Background] Klumpp H, Amir N. Examination of vigilance and disengagement of threat in social anxiety with a probe detection task. Anxiety Stress Coping. 2009 May;22(3):283-96. doi: 10.1080/10615800802449602. PMID 19253172
- [Background] Sportel BE, de Hullu E, de Jong PJ, Nauta MH. Cognitive bias modification versus CBT in reducing adolescent social anxiety: a randomized controlled trial. PLoS One. 2013 May 14;8(5):e64355. doi: 10.1371/journal.pone.0064355. Print 2013. PMID 23691203
- [Background] Beard C, Weisberg RB, Amir N. Combined cognitive bias modification treatment for social anxiety disorder: a pilot trial. Depress Anxiety. 2011 Nov;28(11):981-8. doi: 10.1002/da.20873. Epub 2011 Sep 2. PMID 21898705
- [Background] Emmelkamp PM. Attention bias modification: the Emperor's new suit? BMC Med. 2012 Jun 25;10:63. doi: 10.1186/1741-7015-10-63. PMID 22731990
- [Background] Merikangas KR, He JP, Burstein M, Swanson SA, Avenevoli S, Cui L, Benjet C, Georgiades K, Swendsen J. Lifetime prevalence of mental disorders in U.S. adolescents: results from the National Comorbidity Survey Replication--Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):980-9. doi: 10.1016/j.jaac.2010.05.017. Epub 2010 Jul 31. PMID 20855043
- [Background] Carleton RN, McCreary DR, Norton PJ, Asmundson GJ. Brief fear of negative evaluation scale-revised. Depress Anxiety. 2006;23(5):297-303. doi: 10.1002/da.20142. PMID 16688736
- [Background] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Background] Crocetti E, Hale WW 3rd, Fermani A, Raaijmakers Q, Meeus W. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED) in the general Italian adolescent population: a validation and a comparison between Italy and The Netherlands. J Anxiety Disord. 2009 Aug;23(6):824-9. doi: 10.1016/j.janxdis.2009.04.003. Epub 2009 Apr 23. PMID 19427168
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Tottenham N, Tanaka JW, Leon AC, McCarry T, Nurse M, Hare TA, Marcus DJ, Westerlund A, Casey BJ, Nelson C. The NimStim set of facial expressions: judgments from untrained research participants. Psychiatry Res. 2009 Aug 15;168(3):242-9. doi: 10.1016/j.psychres.2008.05.006. Epub 2009 Jun 28. PMID 19564050
- [Background] Mathyssek CM, Olino TM, Hartman CA, Ormel J, Verhulst FC, Van Oort FV. Does the Revised Child Anxiety and Depression Scale (RCADS) measure anxiety symptoms consistently across adolescence? The TRAILS study. Int J Methods Psychiatr Res. 2013 Mar;22(1):27-35. doi: 10.1002/mpr.1380. Epub 2013 Mar 11. PMID 23483654
- [Background] Inderbitzen-Nolan H, Davies CA, McKeon ND. Investigating the construct validity of the SPAI-C: comparing the sensitivity and specificity of the SPAI-C and the SAS-A. J Anxiety Disord. 2004;18(4):547-60. doi: 10.1016/S0887-6185(03)00042-2. PMID 15149713
- [Background] EU Commission. Toolkit Gender in EU-funded research. Luxembourg, Publications Office of the European Union, 2007.
- [Background] Beidel DC, Turner SM, Morris The Social Phobia and Anxiety Inventory for Children (SPAI-C). Toronto, ON, Multi-Health Systems, 1998.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 2,900 students were invited to take part through Irish second-level schools. N=545 provided assent and parental consent. N=12 were excluded based on exclusion criteria and N=36 were absent for screening.
  N=497 completed screening of which N=130 met the inclusion criteria. Data were collected between September 2014 and May 2015.
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 64 | 66
Completed | 59 | 61
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Missed Post-intervention Data Collection | 2 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Comparison of baseline data for participants who completed the intervention/placebo training.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 61 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.97 (.74) | 15.93 (.68) | 15.95 (.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 23 | 27 | 50
Region of Enrollment [Number; unit: participants]
  Ireland | 59 | 61 | 120
Previously Used Mental Health Services [Number; unit: participants] — Participants answered the following question:
  Have you used any of the following services? Mental health drop in services, Mental health apps (applications), Online support groups (One-on-one support or Support forum), E-mail support services, Helplines
  participants
    Yes | 13 | 8 | 21
    No | 46 | 53 | 99
Threat Bias Measurement [Mean (Standard Deviation); unit: milliseconds] — The threat bias measurement consisted of 120 trials of the dot-probe task, 80 of which contained angry-neutral face pairs and 40 of which contained neutral-neutral face pairs. The threat bias score equal the mean of neutral NT trials minus mean of threat NT trials. A threat bias scores >0 indicate a bias towards threat, whereas scores <0 mean that the participant is slower to respond to threatening stimuli than neutral stimuli. Reaction times were measured in milliseconds.
  milliseconds | 4.01 (28.35) | -.06 (19.03) | 1.94 (24.05)
Social Phobia and Anxiety [Mean (Standard Deviation); unit: units on a scale] — Measured using the Social Phobia and Anxiety Inventory for Children (SPAI-C; Beidel et al., 1998, 2000).
  The Social Phobia and Anxiety Inventory for Children (SPAI-C). The SPAI-C (Beidel et al., 1998, 2000) is a 26-item, self-report measure exploring anxiety in social situations. Responses are indicated using a 3-point Likert scale from 0 = never or hardly ever to 2 = most of the time or always with scores ranging from 0-52. Higher scores on the SPAI-C represent higher levels of social anxiety.
  units on a scale | 29.15 (7.47) | 31.49 (7.53) | 30.34 (7.56)
Fear of Negative Evaluation [Mean (Standard Deviation); unit: units on a scale] — Measured using the Brief Fear of Negative Evaluation-Revised (BFNE-R; Carleton et al., 2006).
  The BFNE-R (Carleton, McCreary, Norton, & Asmundson, 2006) is a 12-item, revised version of the BFNE (Leary, 1983) used to elicit respondents' fear of negative evaluation. Responses are indicated using a 5-point Likert scale response format from 0 = not at all characteristics of me to 4 = entirely characteristic of me. Scores range from 0 to 48. Higher scores indicate higher fear of negative evaluation.
  units on a scale | 31.29 (10.38) | 31.80 (9.67) | 31.55 (9.99)
Anxiety Related Disorders [Mean (Standard Deviation); unit: units on a scale] — The Screen for Child Anxiety Related Emotional Disorders (SCARED)(Birmaher et al., 1997) is a 41-item measure which has five subscales. Responses use a 3-point Likert scale, 0 = not true, or hardly ever true to 2 = very true or often true. The subscales are: Generalized Anxiety Disorder (GAD) (9 items, range 0-18); Panic Disorder (13 items, 0-26); Separation Anxiety Disorder (8 items, 0-16); and Social Phobia (7 items, 0-14), and School Avoidance (4 items, 0-8). Subscales are summed to provide a total score (range 0-82; while scores over 25 may be indicative of an anxiety disorder).
  units on a scale | 36.05 (12.31) | 39.46 (13.81) | 37.78 (13.15)
Depression Symptoms [Mean (Standard Deviation); unit: units on a scale] — The Revised Child Anxiety and Depression Scale - Major Depressive Disorder (RCADS-MDD). The major depressive disorder subscale of the RCADS (Chorpita, Yim, Moffitt, Umemoto, & Francis, 2000) is a 10-item subscale exploring symptoms of MDD as characterised by the DSM-IV, with on a 4-point Likert scale ranging from 0 = never to 3 = always. Scores range from 0 to 30. A score of 11 or higher has been shown to optimise sensitivity and specificity for the prediction of MDD (Ebesutani et al., 2012).
  units on a scale | 11.64 (5.99) | 12.84 (7.31) | 12.25 (6.69)

OUTCOME MEASURES:

1. Primary Outcome: Threat Bias Measurement at 4-week Post-intervention and 12-week Follow-up
Description: The bias measurement protocol consists of 120 trials (80 angry-neutral and 40 neutral-neutral presentations). Angry face location, probe location, probe type and actor are all fully counterbalanced in presentation. The participant must perform with more than 70% accuracy on the first 10 trials.The threat bias measurement consisted of 120 trials of the dot-probe task, 80 of which contained angry-neutral face pairs and 40 of which contained neutral-neutral face pairs. The threat bias score equal the mean of neutral NT trials minus mean of threat NT trials. A threat bias scores >0 indicate a bias towards threat, whereas scores <0 mean that the participant is slower to respond to threatening stimuli than neutral stimuli. Reaction times were measured in milliseconds.
Time Frame: Post-intervention (week 4), and 12-week follow-up
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 59 | 61
milliseconds
  Post-intervention | 1.77 (17.65) | 1.72 (17.07)
  Follow-up | 1.17 (15.94) | 2.27 (18.29)
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority or Other; p > .05, ANOVA — Group x Time interaction p-value: >.05; Gender p-value: >.05; 2x2x3 repeated measures ANOVA. 2 between-subjects factors (Group; Gender) and 1 within-subject factor (Time). P value adjusted to p < .025

2. Primary Outcome: Social Phobia and Anxiety at 4-week Post-intervention and 12-week Follow-up
Description: The Social Phobia and Anxiety Inventory for Children (SPAI-C)(Beidel et al., 1998, 2000) is a 26-item, self-report measure exploring anxiety in social situations. Responses are indicated using a 3-point Likert scale from 0 = never or hardly ever to 2 = most of the time or always with scores ranging from 0-52. Higher scores on the SPAI-C represent higher levels of social anxiety.
Time Frame: Post-intervention (week 4), and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 59 | 61
units on a scale
  Post-intervention | 29.24 (7.89) | 30.67 (8.22)
  Follow-up | 27.12 (8.89) | 29.74 (9.10)
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority or Other; p > .05, ANOVA — Group x Time interaction p-value: >.05; Gender p-value: =.026; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Fear of Negative Evaluation at 4-week Post-Intervention and 12-week Follow-Up
Description: A 12-item self-report questionnaire to measure fear of negative evaluation - Brief Fear of Negative Evaluation Questionnaire -II (BFNE-II; Carleton et al., 2007). The BFNE-R (Carleton, McCreary, Norton, & Asmundson, 2006) is a 12-item, revised version of the BFNE (Leary, 1983) used to elicit respondents' fear of negative evaluation. Responses are indicated using a 5-point Likert scale response format from 0 = not at all characteristics of me to 4 = entirely characteristic of me. Scores range from 0 to 48. Higher scores indicate higher fear of negative evaluation
Time Frame: Post-intervention (week 4), and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 59 | 61
units on a scale
  Post-intervention | 32.73 (13.72) | 31.5 (10.88)
  Follow-up | 31.36 (11.83) | 30.6 (11.21)
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority or Other; p > .05, ANOVA — Group x Time interaction p-value: >.05; Gender p-value: >.05; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Anxiety Related Disorders at 4-week Post-intervention and 12-week Follow-up
Description: The Screen for Child Anxiety Related Emotional Disorders (SCARED)(Birmaher et al., 1997) is a 41-item measure which has five subscales. Responses use a 3-point Likert scale, 0 = not true, or hardly ever true to 2 = very true or often true. The subscales are: Generalized Anxiety Disorder (GAD) (9 items, range 0-18); Panic Disorder (13 items, 0-26); Separation Anxiety Disorder (8 items, 0-16); and Social Phobia (7 items, 0-14), and School Avoidance (4 items, 0-8). Subscales are summed to provide a total score (range 0-82; while scores over 25 may be indicative of an anxiety disorder).
Time Frame: Post-intervention (week 4), and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 59 | 61
units on a scale
  Post-intervention | 35.05 (13.95) | 37.49 (14.37)
  Follow-up | 33.71 (14.78) | 35.41 (14.59)
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority or Other; p > .05, ANOVA — Group x Time interaction p-value: >.05; Gender p-value: <.0001; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Depression Symptoms at 4-week Post-intervention and 12-week Follow-up
Description: The Revised Child Anxiety and Depression Scale - Major Depressive Disorder (RCADS-MDD). The major depressive disorder subscale of the RCADS (Chorpita, Yim, Moffitt, Umemoto, & Francis, 2000) is a 10-item subscale exploring symptoms of MDD as characterised by the DSM-IV, with on a 4-point Likert scale ranging from 0 = never to 3 = always. Scores range from 0 to 30. A score of 11 or higher has been shown to optimise sensitivity and specificity for the prediction of MDD (Ebesutani et al., 2012).
Time Frame: Post-intervention (week 4), and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 59 | 61
units on a scale
  Post-intervention | 12.71 (6.23) | 13.30 (7.78)
  Follow-up | 11.88 (6.86) | 12.57 (7.76)
Statistical Analysis 1: Comparison: Placebo vs Intervention; Test type: Superiority or Other; p > .05, ANOVA — Group x Time interaction p-value: >.05; Gender p-value: =.007; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Placebo | Intervention
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66
Other Adverse Events (participants affected / at risk) | 0/64 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No